CLINICAL TRIAL: NCT05700500
Title: Long-term Treatment of Calcifying Tendinopathy of the Shoulder With Focused Shock Waves or Ultrasound-Guided Needling and Lavage: a Randomized Clinical Trial
Brief Title: Comparison of Focused Shock Waves or Ultrasound-Guided Needling and Lavage in Patients With Calcifying Tendinopathy of the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC123-19_FJD
Record Dates: First submitted 2022-10-10; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Calcific Tendinopathy of Shoulders; Extracorporeal Shockwave Therapy; Ultrasound Guided Barbotage Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- shockwave therapy (Experimental): The calcification will be located by ultrasound and the energy will be applied in the precise place. 3 sessions will be carried out as follows: 1, 2, 3 weeks This procedure will be carried out by a single experienced Physical and Rehabilitation medical doctor
  Interventions: Procedure: shockwave therapy, barbotage and infiltration
- Ultrasound-Guided Barbotage (Experimental): The calcification will be located by ultrasound. By injecting serum at high pressure, it is intended to wash away the calcification. A subacromial inyection will be associated with this procedure. A maximum of 3 Ultrasound-Guided Barbotage will be performed with an interval of 6 weeks between each puncture. This procedure will be performed by two experienced radiologists
  Interventions: Procedure: shockwave therapy, barbotage and infiltration
- us guided subacromial injections (Experimental): An US guided subacromial injection (1 cc of corticostheroid ) and anesthetic (2 cc of mepivacaine) will be performed. The periodicity will be one infiltration every 8-10 weeks, being able to carry out a maximum of 3 per year.
  Interventions: Procedure: shockwave therapy, barbotage and infiltration

INTERVENTIONS:
Procedure: shockwave therapy, barbotage and infiltration — ultrasound guided interventions

SUMMARY:
Currently, the only study comparing the long-term results of these procedures (two years) is that of Kim.(24) This study is the first randomized, blinded clinical trial comparing ultrasound-guided percutaneous lavage ( UPL) for rotator cuff calcific tendinopathy with subacromial injection vs. Shock (1000 impulses/0.36mJ/mm2), obtaining clinical improvement and reabsorption of calcification in both groups. In this study, greater effectiveness was observed in terms of pain improvement and functional recovery in these patients in the short term than in those undergoing UPL: The results of this study were obtained through radiographic evaluation (AP X-ray of the shoulder) before and after intervention and clinical evaluation in both groups using the scales of the American Society of Shoulder and Elbow Surgeons (ASES), the Simple Shoulder Test (SST) and the Visual Analogue Scale (VAS).

Our future work may add many interesting data to the comparative study of these two techniques, since it would provide new results, overcoming the limitations of the only similar study in the literature today.

On the one hand, the radiological selection of patients will be carried out with shoulder X-rays and a shoulder ultrasound performed by two expert musculoskeletal radiologists from this center and validated by interobserver correlation. This will allow a detailed selection of patients according to the characteristics and phases of the calcification that they present. Sonographically, calcifications are classified into three types (according to Garner's 1993 classification): type I, II and III. As we have previously mentioned, calcific tendinopathy is a self-limited disease and we know that calcifications in phase III or in the resorption phase tend to resolve spontaneously. The control ultrasound that will be performed on the patients will also be performed by the same expert musculoskeletal radiologists who have performed the interobserver correlation study.

Secondly , we are going to define a maximum number as well as the exact protocol for carrying out the Eco - guided Puncture Lavage technique .

Another contribution of our work is that we will carry out an evaluation of the differences between both techniques up to two years post-treatment, which will allow us to know the long-term evolution of the results.

ELIGIBILITY:
Inclusion criteria.

* Patients over 18 years of age
* Patients who agree to participate in the study and provide written Informed Consent
* Complete shoulder mobility.
* No associated cervicobrachialgia or associated shoulder injuries.
* No previous shoulder interventions.
* Calcification stage I-II according to the Gartner scale (diagnosed by AP X-ray of the shoulder and ultrasound that will be performed by two radiologists who are experts in musculoskeletal)
* Calcium greater than 0.5 cm
* Pain clinic (VAS > 5) of more than three months of evolution

  • Exclusion criteria
* Pacemakers
* Coagulation disorders
* Pregnancy
* Active neoplastic process.
* Infiltration with corticosteroids less than 6 weeks ago.
* Contraindication to corticosteroid treatment
* Previous treatment with shock waves and / or puncture-aspiration
* Cuff pathology (tear)
* No tolerance to SW
* Previous surgeries on the same shoulder.
* Absolute contraindications for focal shock waves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Results of shoulder function | 3months , 6 months , 1 year

SECONDARY OUTCOMES:
Change in Eva scale to assess the pain | 3months , 6 months , 1 year
  0-10
change in worc scale to assess shoulder function | 3months , 6 months , 1 year
  0-210
changes in Constant scale to assess shoulder function | 3months , 6 months , 1 year
  0-100
rate of complications of the rotator cuff assessed by MRI | 3months , 6 months , 1 year
  bursitis , intraosseous migration , intramuscular migration
changes in EuroQol5d scale to assess the subjective satisfaction of the patient | 3months , 6 months , 1 year
  0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Jimenez Díaz Hospital, Madrid, Spain